CLINICAL TRIAL: NCT02359227
Title: A Study Assessing the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Open-Label, Continuous, Stepwise, Dose Increasing, Subcutaneous Infusion of Cenderitide Via the Insulet Drug Delivery System in Subjects With Stable, Chronic Heart Failure
Brief Title: Safety Study of Cenderitide in Stable Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDNP-578-01
Record Dates: First submitted 2015-02-02; First posted 2015-02-09 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure; Natriuretic Peptides; Cenderitide
MeSH Terms: conditions — Heart Failure | interventions — cenderitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cenderitide (Experimental): Cenderitide will be administered as four, 48-hour, continuous, subcutaneous infusion rates of 0.5, 1.0, 2.0 and 3.0 ng/kg/min totaling up to eight sequential days of dosing.
  Interventions: Drug: Cenderitide

INTERVENTIONS:
Drug: Cenderitide — Cenderitide is a dual receptor natriuretic peptide.

SUMMARY:
Planned enrollment is approximately twelve subjects with stable chronic heart failure. Enrolled subjects will receive up to eight sequential days of continuous, stepwise, dose increasing, subcutaneous (SQ) infusions of open-label cenderitide via the Insulet Drug Delivery System. Planned infusion rates of cenderitide will be administered to subjects continuously during four, 48-hour infusion periods.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, ≥ 18 years of age
* Body Mass Index (BMI) of 18-40 kg/m2, inclusive
* Current or historical New York Heart Association (NYHA) functional class ≥ II
* At least one of the following: documented systolic heart failure with an ejection fraction (EF) ≤ 40% and/or a historical measurement of plasma BNP ≥ 150 pg/mL (or NT-proBNP ≥ 600 pg/mL)
* Systolic blood pressure 100-160 mmHg
* Stable and compliant treatment with oral heart failure medications for at least 4 weeks prior to Screening

Key Exclusion Criteria:

* Known hypersensitivity or allergy to natriuretic peptide or its components, nesiritide, other natriuretic peptides or related compounds
* Current clinical diagnosis of acute decompensated heart failure (ADHF)
* Clinical diagnosis of acute coronary syndrome (ACS) within 30 days prior to Screening.
* Symptomatic postural hypotension
* Evidence of uncorrected volume or sodium ≤ 130 mmol/L or other condition that would predispose the patient to adverse events
* Clinically significant aortic or mitral valve stenosis
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (not including restrictive mitral filling patterns)
* Severe renal failure defined as creatinine clearance < 45 mL/min as estimated by either the Cockcroft-Gault or the MDRD equations
* Significant pulmonary disease (e.g., history of oral daily steroid dependency, history of Carbon Dioxide (CO2) retention or need for intubation for acute exacerbation, or currently receiving IV steroids)
* Known hepatic impairment as indicated by any of the following: A) total bilirubin > 3 mg/dL; B) albumin < 2.8 mg/dL, with other signs or symptoms of hepatic dysfunction; C) increased ammonia levels, if performed, with other signs or symptoms of hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-04-02 (Actual); Study Completion 2015-04-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by changes in vital signs (blood pressure, heart rate, and body temperature), clinical laboratory tests, adverse events, 12-lead ECGs, and physical examinations compared to pre-dose, baseline measurements. | Measurements performed at regular intervals on Days 1-10, and at the safety follow-up visit (Day 16 ± 2 days).
Pharmacokinetic (PK) profile of cenderitide as measured in area under the blood concentration-curve (AUC) from time zero to 48 hours post each infusion rate start, maximum blood concentration (Cmax), and time of maximum blood concentration (Tmax). | PK blood collection at regular intervals on Days 1-10.
Pharmacodynamic (PD) response as assessed by changes in blood pressure, heart rate, weight, fluid balance (intake/output), plasma cGMP, ANP, NT-proBNP, and aldosterone, and urine cGMP compared to pre-dose baseline assessments. | PD assessments performed at regular intervals on Days 1-10, and at the safety follow-up visit (Day 16 ± 2 days).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States